CLINICAL TRIAL: NCT00850148
Title: Comparison of Anwar and Melles Techniques in Deep Anterior Lamellar Keratoplasty (DALK) for Keratoconus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Other Study IDs: 8721
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2009-02

CONDITIONS: Keratoconus
Keywords: Anwar; Melles; Keratoconus
MeSH Terms: conditions — Keratoconus

ARMS (2):
- Melles (Experimental)
  Interventions: Procedure: Melles
- Anwar (Experimental)
  Interventions: Procedure: Anwar

INTERVENTIONS:
Procedure: Anwar — Anwar surgical method
  Arms: Anwar
Procedure: Melles — Melles surgical method
  Arms: Melles

SUMMARY:
This study will be performed on patients who come to labbafinejad ophthalmic clinic from 20 March 2008. Keratoconus diagnosis will be determined by clinical finding in slit lamp, keratometery and topographic characteristics. Patients will be randomly placed in group A and B. In group A, Anwar surgical method and in B, Melles surgical method, will be done. This is not a blind study due to surgeons' knowledge. All patients will receive Btamethazone drop and Chloramphenicol every 6 hours and will be tapered in two months. In the end anatomical results, complications, BCVA, UCVA, astigmatism, endothelial cell numbers will be compared in two groups by using specular microscopy. Contrast sensivity, central corneal diameter, interface wrinkling and opacity will be measured by metrovison, Confoscan, Photoslit in months 3, 6, 12, respectively and will be evaluated afterwards.

ELIGIBILITY:
Inclusion Criteria:

* patients with keratoconus
* 15<age<45
* contact lens intolerance

Exclusion Criteria:

* Having a history of any other ophthalmic or systemic problem
* Central corneal scar
* descemet's membrane detachment

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Ophtalmic Research Centre, Tehran, Tehran Province
  - Farid Karimian,MD, Tehran, Tehran Province